CLINICAL TRIAL: NCT03885804
Title: Efficacy of Perineural Versus Intravenous Dexmedetomidine as an Adjuvant to Quadratus Lamborum Block for Pediatrics Undergoing Laparoscopic Pyeloplasty. A Prospective Randomized Double Blinded Study
Brief Title: Perineural Versus IV Dexmedetomidine as Adjuvant to Quadratus Lamborum Block for Pediatrics Undergoing Pyeloplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Associte professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 06/ 2019
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pain, Postoperative
Keywords: quadratus - dexmedetomidine- bupivavaine- perineural
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomisation by concealed envelope method
Who Masked: Participant, Outcomes Assessor
Masking Description: a physician assessing outcomes blinded to the nature of the study as first and second rescue analgesics respectively.Drug packs will be prepared before commencement of the study by a pharmacist unaware of the nature of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lamborum dexmedetomidine intravenous group (Sham Comparator): Patients will receive quadratus lamborum block on the same surgical side.a bolus of 0.5 ml/Kg bupivacaine 0.25% in addition to 2ml normal saline will be injected then dexmedetomidine (precedex 200 micrograms per 2ml, Abbott laboratories, Abbott park, IL, USA) which will be prepared in concentration 1μg/ml. 1ml/kg loading dose will be given over 10 min followed by 0.5 ml/kg/h infusion maintenance dose till the end of surgery
  Interventions: Drug: Quadratus lamborum dexmedetomidine intravenous
- Quadratus lamborum dexmedetomidine perineural group (Active Comparator): Patients will receive quadratus lamborum block on the same surgical side. Patients will receive perineural dexmedetomidine of 1μ g/kg diluted to 2 mL with 0.9% saline added to 0.5 ml/kg of 0.25% bupivacaine in addition to saline infusion 1ml/kg IV loading dose followed by by 0.5 ml/kg/h infusion maintenance dose till the end of surgery.
  Interventions: Drug: Quadratus lamborum dexmedetomidine perineural group(

INTERVENTIONS:
Drug: Quadratus lamborum dexmedetomidine intravenous — Patients will receive quadratus lamborum block on the same surgical side then a bolus of 0.5 ml/Kg bupivacaine 0.25% in addition to 2ml normal saline will be injected then dexmedetomidine (precedex 200 micrograms per 2ml, Abbott laboratories, Abbott park, IL, USA) which will be prepared in concentration 1μg/ml. 1ml/kg loading dose will be given over 10 min followed by 0.5 ml/kg/h infusion maintenance dose till the end of surgery
  Other Names: (QD IV group)
  Arms: Quadratus lamborum dexmedetomidine intravenous group
Drug: Quadratus lamborum dexmedetomidine perineural group( — Patients will receive quadratus lamborum block on the same surgical side then1μ g/kg diluted to 2 mL with 0.9% saline added to 0.5 ml/kg of 0.25% bupivacaine in addition to saline infusion 1ml/kg IV loading dose followed by by 0.5 ml/kg/h infusion maintenance dose till the end of surgery.
  Other Names: QD PN group
  Arms: Quadratus lamborum dexmedetomidine perineural group

SUMMARY:
this prospective parallel group double blinded study will be conducted over 50 pediatric patients ASA (American Association of Anesthesiologists) I and II between the age of 8-13 years old,who will be scheduled for laparoscopic pyeloplasty.Patients will be randomly allocated into 2 study groups: Quadratus lamborum dexmedetomidine intravenous group(QD IV group) and Quadratus lamborum dexmedetomidine perineural group(QD PN group.Patients in both groups will receive quadratus lamborum block .In QD IV group a bolus of 0.5 ml/Kg bupivacaine 0.25% in addition to 2ml normal saline will be injected then dexmedetomidine.1ml/kg loading dose will be given over 10 min followed by 0.5 ml/kg/h infusion maintenance dose till the end of surgery. In QD PN, patients will receive perineural dexmedetomidine of 1μ g/kg diluted to 2 mL with 0.9% saline added to 0.5 ml/kg of 0.25% bupivacaine in addition to saline infusion 1ml/kg IV loading dose followed by by 0.5 ml/kg/h infusion maintenance dose till the end of surgery.Time to first analgesic requirement ( primary outcome) , Wong-Baker FACES Pain Rating Scale scores will be recorded at 2, 6, 8,12, 18 and 24h postoperatively, the degree of sedation will be assessed by Ramsay sedation scores(fig.2)(9) at the same time points, hemo-dynamics as systolic and diastolic blood pressures and heart rates will be recorded at PACU discharge then 4 hourly, total dose of morphine consumption, , the length of hospital stay, incidence of postoperative complications as hypotension, bradycardia, vomiting, pruritis and respiratory depression

DETAILED DESCRIPTION:
this prospective parallel group double blinded study will be conducted over 50 pediatric patients ASA (American Association of Anesthesiologists) I and II between the age of 8-13 years old, ASA physical status I and II, who will be scheduled for laparoscopic pyeloplasty and performed by the same surgical team. This study will be carried out at Ain Shams University hospitals. Written informed consent will be obtained from the parents. Exclusion criteria will include: History of developmental delay or mental retardation, parent refusal, history of allergic reactions to local anesthetics, rash or infection at the injection site, anatomical abnormality, bleeding disorders, history of cardiac, neurological, impaired renal function defined by s-creatinine >150 μmol/L and impaired hepatic function. Preanesthetic evaluation and routine investigations will be carried out on the night of surgery and patients shall be fasting for 6 hours. After an intravenous (IV) cannula (22G) is secured , and midazolam 0.02 mg/kg iv will be administered to all patients before transfer to the operating room. Standard monitoring devices as ECG, Non- invasive blood pressure, nasopharyngeal temperature probe and pulse oximetry will be placed then baseline systolic and diastolic blood pressures and heart rate will be recorded. Induction of general anesthesia (GA) will be accomplished using propofol 1-2mg/kg, fentanyl will be administered intravenously at 1μg/kg, Intubation will be facilitated by atracurium (0.5 mg/kg) then an appropriately sized endotracheal tube will be placed.All patients will be mechanically ventilated with volume controlled mode with targeted EtCO2 (30-35 mmHg) and anesthesia will be maintained with 1.2% isoflurane in a mixture of 50% air and oxygen in all patients throughout the procedure which will be adjusted according to the adequacy of anesthesia. Intraoperative hypothermia will be prevented by warm intravenous fluids (15 ml/kg lactated ringer solution in the first hour then completed according to fluid chart) and warm mattress.

A total of 50 patients will be randomly allocated into 2 study groups: Quadratus lamborum dexmedetomidine intravenous group(QD IV group) and Quadratus lamborum dexmedetomidine perineural group(QD PN group) using concealed envelope method, physicians assigned participants to interventions according to allocation: Patients in both groups will receive quadratus lamborum block on the same surgical side , first the patients will be placed in the lateral position then turned to supine position after completion of the block. Under aseptic conditions,a high-frequency linear probe (SonoSite HFL50x, 15- 6 MHz, 55-mm broadband linear array) will be placed on the lateral abdomen, between the costal margin and iliac crest. The three abdominal muscles, external oblique (EO), internal oblique (IO), and transversus abdominis muscle (TA), will be identified then the probe will be moved posteriorly and QL muscle (QLM) will visualized. A 22-G block needle (Stimuplex D, Braun, Hongo, Bunkyo-ku,Tokyo) will be oriented in plane, from anterior to posterior direction, and the needle tip will be positioned between the anterior border of QLM and its fascia: In QD IV group a bolus of 0.5 ml/Kg bupivacaine 0.25% in addition to 2ml normal saline will be injected then dexmedetomidine (precedex 200 micrograms per 2ml, Abbott laboratories, Abbott park, IL, USA) which will be prepared in concentration 1μg/ml. 1ml/kg loading dose will be given over 10 min followed by 0.5 ml/kg/h infusion maintenance dose till the end of surgery. In QD PN, patients will receive perineural dexmedetomidine of 1μ g/kg diluted to 2 mL with 0.9% saline added to 0.5 ml/kg of 0.25% bupivacaine in addition to saline infusion 1ml/kg IV loading dose followed by by 0.5 ml/kg/h infusion maintenance dose till the end of surgery. Drug packs will be prepared before commencement of the study by a pharmacist unaware of the nature of the study, after 15 minutes of the block, surgical incision will be allowed but in case of conversion to open surgical procedure (laparotomy) patients will be excluded from the study.The average end-tidal isoflurane, total intraoperative fentanyl dose and incidence of intraoperative complications as hypotension, If the blood pressure dropped more than 30% of the baseline values, it will be managed by 10 ml/kg normal saline and ephedrine injection and/or bradycardia is defined as drop of heart rate more than 20% of the baseline values which will be managed by atropine 0.02mg/kg, all will be recorded. Inadequate analgesia is defined as more than 20% increase in mean blood pressure and heart rate after skin incision and during surgical procedure which will be managed by administration of 0.5 μg/kg fentanyl. At the end of surgical procedure, muscle relaxation will be reversed with neostigmine 50 μg/kg and atropine sulfate 20 μg/kg. Patients will extubated and shifted to the post-anaesthesia care unit.

The recovery time (The elapsed time for the patient to open his eyes upon command after discontinuation of Isoflurane) will be recorded. In postoperative anaesthesia care unit, postoperative monitoring of the hemodynamics will be undergone by a well trained nurse. when pain score >4 on Wong-Baker FACES Pain Rating Scale (8) (fig.1), patients will be given morphine 0.05 mg·kg-1 6 hourly and acetaminophen IV 15mg/kg 6 hourly will be administered by a physician blinded to the nature of the study as first and second rescue analgesics respectively. Time to first analgesic requirement ( primary outcome) , Wong-Baker FACES Pain Rating Scale scores will be recorded at 2, 6, 8,12, 18 and 24h postoperatively, the degree of sedation will be assessed by Ramsay sedation scores(fig.2)(9) at the same time points, hemo-dynamics as systolic and diastolic blood pressures and heart rates will be recorded at PACU discharge then 4 hourly, total dose of morphine consumption, , the length of hospital stay, incidence of postoperative complications as hypotension, bradycardia, vomiting, pruritis and respiratory depression, which is defined as respiratory rate less than 10 breathes/min will be recorded. If the blood pressure dropped more than 30% 0f the baseline values, it will be managed by 10 ml/kg normal saline and ephedrine injection. Bradycardia is defined as drop of heart rate more than 20% of the baseline values. It will be managed by atropine 0.02mg/kg. Attacks of vomiting will be managed by ondansetron 0.1 mg/kg iv.

ELIGIBILITY:
Inclusion Criteria:

* paediatrics
* 8-13 years old
* ASA I-II
* laparoscopic pyeloplasty

Exclusion Criteria:

* developmental delay or mental retardation
* parent refusal
* history of allergic reactions to local anesthetics
* infection at the injection site bleeding disorders history of cardiac, neurological, impaired renal function defined by s-creatinine >150 μmol/L

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine consumption | 24 hours
  mg/kg

SECONDARY OUTCOMES:
recovery time | 15-24 minutes
  The elapsed time for the patient to open his eyes upon command after discontinuation of Isoflurane
Ramsay sedation scores | 24 hours postoperative
  Ramsay Sedation Scale
  1 Anxious or restless or both Unacceptable; increase sedation 2 Cooperative, orientated and tranquil Acceptable; no action necessary 3 Responding to commands Acceptable; no action necessary 4 Brisk response to stimulus Acceptable; no action necessary 5 Sluggish response to stimulus Unacceptable; monitor respiratory status and sedation level until stable at 2 or 3 6 No response to stimulus Unacceptable; monitor respiratory status and sedation level until stable at 2 or 3
incidence of postoperative complications | 24 hours postoperative
  Mann Witney test

CONTACTS AND LOCATIONS:
Overall Officials: Reem Elkabarity, Study Chair — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after discussion with other authors, the study protocol, statistical analysis and informed consent will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 4-6 months
Access Criteria: The collected data will be coded, tabulated, and statistically analysed using PASS program setting alpha error at 5% and power at 95%,.
  Descriptive statistics will be carried out for numerical parametric data and presented as mean±SD, whereas categorical data will be presented as number and percentage. Variables such as demographic data and comorbidities will be compared using the χ2-test. A P value less than 0.05 will be considered significant Requests will be reviewed by authors